CLINICAL TRIAL: NCT06292182
Title: Can Red Light Lift Droopy Eyelids? An Open-label Proof-of-concept Study
Brief Title: Red Light Ptosis Proof-of-Concept
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160802; 332942 (Other: IRAS); 58964 (Other: CPMS)
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Mitochondrial Diseases; Blepharoptosis
MeSH Terms: conditions — Mitochondrial Diseases; Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment start at baseline (Experimental)
  Interventions: Device: Near-infrared light
- Delayed treatment start at 3 months from baseline (Experimental)
  Interventions: Device: Near-infrared light

INTERVENTIONS:
Device: Near-infrared light — daily application of near-infrared light

SUMMARY:
This study tests a new treatment to help with droopy eyelids (ptosis) and eye movement problems (squint) in children and young people with genetically confirmed mitochondrial conditions - using red-light.

We use a torch to shine a red light through the closed eyelid for 3 minutes a day. The study will run for 18 months.

We believe that this treatment could help strengthen the muscle in the eyelid to make it easier to open the eyes, and could also help some children with squint.

ELIGIBILITY:
Inclusion: Age 3 to less than 18 years Genetically confirmed diagnosis of primary mitochondrial disease (known pathogenic mutation(s) in mitochondrial or nuclear DNA known to cause primary mitochondrial disease) Ptosis

Exclusion: Genetic diagnosis not consistent with primary mitochondrial disease. No genetic diagnosis Unable to cooperate with light treatment or ophthalmological assessments.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Palpebral fissure width | 3 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No